CLINICAL TRIAL: NCT07209384
Title: CLINICAL EFFICACY OF TRANSARTERIAL CHEMOEMBOLIZATION IN ELDERLY PATIENTS WITH ADVANCED UNRESECTABLE COLORECTAL CANCER
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Junpeng Wang (Other)
Collaborators: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor-Investigator, Junpeng Wang, Chief physician, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Organization: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-10-01
Record Dates: First submitted 2025-10-01; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Unresectable Colorectal Cancer; Advanced Malignancy; Elderly (People Aged 65 or More)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- transarterial chemoembolization with FOLFOX plus/minus intravenous cetuximab/bevacizumab (Experimental)
  Interventions: Procedure: Transarterial chemoembolization

INTERVENTIONS:
Procedure: Transarterial chemoembolization — Transarterial chemoembolization with FOLFOX plus/minus intravenous cetuximab/bevacizumab

SUMMARY:
We plan to conduct a prospective, two-arm, open-label phase Ⅱ study to evaluate whether transarterial chemoembolization with FOLFOX plus/minus intravenous cetuximab/bevacizumab significantly improves the efficacy and safety compared with systemic FOLFOX therapy plus/minus cetuximab/bevacizumab in elderly patients with advanced unresectable colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years, gender not restricted Pathologically confirmed advanced colorectal cancer without the opportunity for curative surgery Karnofsky Performance Status (KPS) score ≥ 60, with an estimated survival time ≥ 3 months At least 1 measurable colorectal lesion No prior systemic chemotherapy, or a minimum interval of 6 months between the last chemotherapy and study enrollment Voluntary signing of the informed consent form

Exclusion Criteria:

* Concomitant other malignant tumors Presence of gastrointestinal perforation Severe cardiovascular and cerebrovascular diseases Patients with hypersensitivity to study drugs or psychiatric disorders

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate；Disease Control Rate | 24 weeks

IPD SHARING:
Plan to Share IPD: Yes